CLINICAL TRIAL: NCT03401333
Title: Feasibility of Augmenting Brief Interventions With Text Messaging to Reduce Adolescent Alcohol and Marijuana Use
Brief Title: Brief Interventions With Text Messaging to Reduce Adolescent Alcohol and Marijuana Use
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000021254
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Alcohol Drinking; Marijuana
MeSH Terms: conditions — Alcohol Drinking; Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: A brief motivational interview and four weeks of text messaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text messaging and brief intervention (Experimental): Brief motivational interview and 4-weeks of text messaging.
  Interventions: Behavioral: Text Messaging and Brief Negotiation Interview

INTERVENTIONS:
Behavioral: Text Messaging and Brief Negotiation Interview — An in-person brief motivational intervention coupled with 4 weeks of motivational text messages

SUMMARY:
This study tests the feasibility of an intervention to prevent risky alcohol or marijuana use that adds a 4-week course of tailored text messaging to a brief motivational intervention for 13-18-year-old adolescents.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 18 years old
* Able to provide consent or assent and parental permission
* have a functioning cell phone without pay-as-you-go text messaging

Exclusion Criteria:

* currently enrolled in any substance abuse program;
* have medical/psychiatric condition that precludes participation

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Enrollment | Baseline
  Number of participants per month that enroll in the study
Retention | 4 weeks
  % of enrolled participants that complete the 4-week follow up assessments
Satisfaction | 4 weeks
  Participant's rating of how much they like the intervention (Likert scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared